CLINICAL TRIAL: NCT01012661
Title: Evaluation of Pain With the Use of Lidocaine-Mixed Radiesse® Injectable Dermal Filler for the Treatment of Nasolabial Folds
Brief Title: Evaluation of Pain With Lidocaine-Mixed Radiesse® Injectable Dermal Filler
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0408329
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Results first posted 2010-01-15 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Nasolabial Folds
Keywords: Moderate to severe wrinkles and folds such as nasolabial folds

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiesse® Mixed with Lidocaine (Experimental): Injectable Dermal Filler. The same 50 participants received both the treatment device and the control device at the same time (left and right sides of face).
  Interventions: Device: Radiesse® Injectable Dermal Filler Mixed with Lidocaine
- Radiesse® without Lidocaine (Active Comparator): Injectable Dermal Filler. The same 50 participants received both the treatment device and the control device at the same time (left and right sides of face.
  Interventions: Device: Radiesse® Injectable Dermal Filler without Lidocaine

INTERVENTIONS:
Device: Radiesse® Injectable Dermal Filler Mixed with Lidocaine — Calcium hydroxylapatite particles suspended in an aqueous based gel carrier mixed with 2% lidocaine hydrochloride (HCl)
  Arms: Radiesse® Mixed with Lidocaine
Device: Radiesse® Injectable Dermal Filler without Lidocaine — Calcium hydroxylapatite particles suspended in an aqueous based gel carrier without 2% lidocaine hydrochloride (HCl)
  Arms: Radiesse® without Lidocaine

SUMMARY:
To assess pain during nasolabial fold treatment using Radiesse® Injectable Dermal Filler mixed with lidocaine.

DETAILED DESCRIPTION:
To assess pain immediately after nasolabial fold treatment with Radiesse® Injectable Dermal Filler mixed with lidocaine in one nasolabial fold compared to Radiesse® Injectable Dermal Filler without lidocaine in the contralateral nasolabial fold.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age.
* Is a candidate for nasolabial fold treatment using Radiesse.
* Understands and accepts the obligation not to receive any other facial procedures in the lower half of the face for 1 month.
* Understands and accepts the obligation to present for all scheduled follow-up visits and is logistically able to meet all study requirements.
* Has approximately symmetrical nasolabial folds.

Exclusion Criteria:

* Has received any type of treatment or procedures including surgery in the nasolabial folds.
* Has received neurotoxins in the lower half of the face in the past 6 months.
* Has received hyaluronic acid, calcium hydroxylapatite (CaHA) or collagen injections in the lower half of the face within past 1 ½ years.
* Has received polylactic acid, polymethyl methacrylate (PMMA), silicone or any other permanent filler in the lower half of the face.
* Has nasolabial folds that are too severe to be corrected in one treatment session.
* Has a history of chronic or recurrent infection or inflammation that would preclude participation in the study.
* Has a known bleeding disorder or is receiving medication that will likely increase the risk of bleeding.
* Is female and of child bearing potential and is pregnant or not using acceptable method of birth control.
* Has had any history of hypersensitivity to Lidocaine or anesthetics of the amide type.
* Has a history of anaphylaxis or multiple severe allergies.
* Has received any investigational product within 30 days prior to study enrollment or is planning to participate in another investigation during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rockville, Maryland
  - New York, New York

REFERENCES:
- [Result] Marmur E, Green L, Busso M. Controlled, randomized study of pain levels in subjects treated with calcium hydroxylapatite premixed with lidocaine for correction of nasolabial folds. Dermatol Surg. 2010 Mar;36(3):309-15. doi: 10.1111/j.1524-4725.2009.01435.x. Epub 2010 Jan 19. PMID 20100272

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiesse® Mixed With Lidocaine & Radiesse® Without Lidocaine: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier containing 2% lidocaine hydrochloride (HCl) and Calcium hydroxylapatite particles suspended in an aqueous based gel carrier without 2% lidocaine hydrochloride (HCl). The same 50 participants received both the treatment device and the control device at the same time (left and right sides of face).
Period: Overall Study
Arm/Group | Radiesse® Mixed With Lidocaine & Radiesse® Without Lidocaine
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier containing 2% lidocaine hydrochloride (HCl) and Calcium hydroxylapatite particles suspended in an aqueous based gel carrier without 2% lidocaine hydrochloride (HCl)
Arm/Group | Radiesse® Mixed With Lidocaine and Radiesse® Without Lidocaine
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Using a 10-cm Visual Analog Pain Scale (1 = no Pain, 10 = Very Severe Pain)
Description: Assessment of difference in pain score in the Radiesse Dermal Filler Mixed with Lidocaine nasolabial fold v. the Radiesse Dermal Filler without Lidocaine nasolabial fold using a 10-cm visual analog pain scale (1 = no pain, 10 = very severe pain).
Time Frame: Immediately after injection (Time 0)
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Radiesse® Mixed With Lidocaine: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier containing 2% lidocaine hydrochloride (HCl)
- Radiesse® Without Lidocaine: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier without 2% lidocaine hydrochloride (HCl)
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 50 | 50
cm | 2.8 (1.9) | 6.6 (2.2)

2. Primary Outcome: Patients With Clinically Significant Reduction in Pain
Description: Assessment of clinical significance of pain reduction in the Radiesse Injectable Dermal Filler Mixed with Lidocaine nasolabial fold v. Radiesse Injectable Dermal Filler without Lidocaine nasolabial fold defined as number of participants with >/= 2cm difference on a visual analog pain scale (1 = no pain, 10 = very severe pain).
Time Frame: Immediately after injection (Time 0)
Measure: Number; unit: Participants
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Number analyzed (Participants) | 50 | 50
Participants | 45 | 0

ADVERSE EVENTS:
Arm/Group | Radiesse® Mixed With Lidocaine | Radiesse® Without Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 46/50 | 45/50
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiesse® Mixed With Lidocaine (N=50) | Radiesse® Without Lidocaine (N=50)
Bruising (Skin and subcutaneous tissue disorders) | 25 (26) | 25 (25)
Itching (Skin and subcutaneous tissue disorders) | 10 (13) | 12 (16)
Pain (Skin and subcutaneous tissue disorders) | 21 (22) | 23 (25)
Redness (Skin and subcutaneous tissue disorders) | 28 (29) | 30 (32)
Swelling (Skin and subcutaneous tissue disorders) | 44 (47) | 42 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves right to review/comment on any manuscript for publication/presentation presenting data from the trial. No manuscript may be submitted for publication without prior review. Investigator agrees to accommodate reasonable requests to protect propriety rights/interests. Investigator must ensure accuracy of results. Investigator shall grant Sponsor right to reproduce/translate/use all copyrighted material from study publications.